CLINICAL TRIAL: NCT05804929
Title: Study on the Phenotype and Gut Microbiome Composition of Healthy Superlean Individuals (BMI < 18.5)
Brief Title: Phenotypic Characteristics of Superlean Individuals Including Gut Microbiome
Status: Completed | Type: Observational
Sponsor: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, John R. Speakman, Professor, Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Other Study IDs: SIAT-IRB-221115-H0628
Record Dates: First submitted 2023-02-17; First posted 2023-04-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Thinness; Health Behavior
Keywords: Superlean; Metabolism; Microbiome; body composition; food intake; food preference
MeSH Terms: conditions — Thinness; Health Behavior; Food Preferences | interventions — Observation; Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Microbial DNA was extracted from frozen fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: 21.5≤BMI<25, age between 25-40 years old, 200subjects.
  Interventions: Other: Observation without intervention
- Superlean: BMI≤18.5, age between 25-40 years old, 200 subjects.
  Interventions: Other: Observation without intervention

INTERVENTIONS:
Other: Observation without intervention — Observation of food intake, body composition, microbiota, genetics, metabolic rate, metabolomics.

SUMMARY:
The goal of this observational study is to build on our previous work to further characterise the phenotype of superlean individuals (BMI < 18.5) when compared to normal BMI people (BMI 21.5 to 25). This will include characterising the body composition, food intake behaviour, circulating hormone levels, genetics and characteristics of the gut microbiota. The investigators expect to recruit up to 200 healthy superlean and control volunteers respectively,

DETAILED DESCRIPTION:
The focus of this work is to characterise the phenotype and genotype of individuals who have low BMI ( < 18.5) but are otherwise healthy and do not have eating disorders. The investigators term this group 'superlean' individuals. The study is observational and the investigators aim to establish a healthy superlean cohort,and use the combined metagenomic and metabolomic multi-omics analysis techniques, combined with imaging and physiological measurements, to focus on the correlation between gut microbiota characteristics and metabolism in superlean population. The investigators expect to recruit up to 200 healthy superlean and control volunteers (BMI 21.5 to 25) respectively, to explore the microbiota characteristics and differences between control and healthy superlean populations by measuring the basic physical indicators and metabolic parameters. This will include analyzing the postprandial hormonal changes, appetite differences, and changes in the gut microbiome and serum metabolome in the two groups of volunteers, establishing the relationship between the gut microbiota and the metabolite and metabolic phenotypes of the body, and exploring the gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Control group (21.5≤ BMI<25), Superlean group (BMI≤18.5)
* Age between 25-40 years old

Exclusion Criteria:

* Having metabolic diseases or eating disorders
* Recent weight loss due to various disease causes
* Being treated for weight loss
* Having an infectious disease
* Pregnant and lactating women
* People with blood sickness, pathological hypo- or hypertension
* People suffering from claustrophobia
* No metal implants in the body
* Use of antibiotics, probiotics, oral laxatives, etc. within 8 weeks

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants are healthy, with no metabolic disorder, 25 - 40 years old
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Weight | Through study completion, an average of 2 years, will be measured on arrival.
  Volunteers will be asked to fast for 10 hours and measured fasting weight.
Height | Through study completion, an average of 2 years, will be measured on arrival.
  Height will be measured by seca 217 stable stadiometer.
Waist circumferences | Through study completion, an average of 2 years, will be measured on arrival.
  Waist circumferences will be measured using a whole body laser scanner.
Hip circumferences | Through study completion, an average of 2 years, will be measured on arrival.
  Hip circumferences will be measured using a whole body laser scanner.
Bone mineral density | Through study completion, an average of 2 years, will be measured on arrival.
  Bone mineral density will be measured by Dual Energy X-ray Absorptiometry (Horizon Wi).
Fat mass | Through study completion, an average of 2 years, will be measured on arrival.
  Fat mass will be measured by Magnetic Resonance Imaging (Shanghai united imaging, uMR 790 ).
Fat free mass | Through study completion, an average of 2 years, will be measured on arrival.
  Fat free mass will be measured by Bioimpedance Analysis (Tanita, MC-980).
Blood pressure | Through study completion, an average of 2 years, will be measured on arrival.
  Systolic and diastolic blood pressure will be measured using an Omron sphygmomanometer.
Glucose | Through study completion, an average of 2 years, will be recorded for a consecutive of 7 days.
  Fasting and post-prandial glucose after a standard meal will be recorded by the continuous glucose monitoring system.
Body temperature | Through study completion, an average of 2 years, will be measured before and after feeding.
  Body temperature will be measured before and after feeding using a thermal imaging camera.
Resting energy expenditure | Through study completion, an average of 2 years, will be measured on arrival.
  The measurement of resting energy expenditure will be performed using indirect calorimetry.
Physical activity | Through study completion, an average of 2 years, will be recorded for a consecutive of 7 days.
  Physical activity of the participants will be recorded using GT3X monitor for a consecutive of 7 days.
Body shape | Through study completion, an average of 2 years, will be measured on arrival.
  Body shape will be measured using a whole body laser scanner.
Energy intake | Through study completion, an average of 2 years, will be measured on arrival.
  Response on standard feeding table, the food consumption will be recorded continuously by balances underneath each food dish. The total energy intake will be calculated in KJ (kilojoule).
Circulating hormones | Through study completion, an average of 2 years, will be measured after standard intervention meal.
  Levels of circulating hormones (including leptin, insulin, ghrelin etc) will be measured when fasted and after a standard intervention meal. Levels of circulating hormones in the serum will be measured by ELISA (Bio Tek, Synergy4) in mmol/L.
Microbiome | Through study completion, an average of 2 years, will be measured after samples collected.
  Abundance of gut microbiome will be from Metagenomic profiling of feces by Illumina.
Metabolites | Through study completion, an average of 2 years, will be measured after samples collected.
  Abundance of metabolites will be from metabolomic profiling of serum and feces by LC-MS (liquid chromatography-mass spectrometry).
Genetics | Through study completion, an average of 2 years, will be measured after samples collected.
  Polymorphic variation will be assessed in a panel of SNPs (single nucleotide polymorphism) previously linked to body composition and physical activity using a Mass array sequencer.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Institute of Advanced Technology,, Shenzhen, China

IPD SHARING:
Plan to Share IPD: No